CLINICAL TRIAL: NCT00332176
Title: A Phase II Randomized, Active-Controlled Study to Assess the Safety, Antiviral Effect, and Pharmacokinetics of Celgosivir in Combination With Peginterferon Alfa-2b and Ribavirin Over 12 Weeks in Treatment-Naïve Patients With Chronic Hepatitis C
Brief Title: A Study to Evaluate the Safety, Antiviral Effect, and Pharmacokinetics of Celgosivir in Combination With Peginterferon Alfa-2b and Ribavirin in Treatment-Naïve Patients With Chronic Hepatitis C
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BioWest Therapeutics Inc (Industry)
Responsible Party: Jim Pankovich, Study Director, MIGENIX Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV-06-001
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2008-04

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Celgosivir; HCV; Genotype 1; Treatment-naive; Early viral kinetics
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — celgosivir; peginterferon alfa-2b; Ribavirin

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Celgosivir
- 2 (Experimental)
  Interventions: Drug: Celgosivir
- 3 (Active Comparator)
  Interventions: Drug: Peginterferon alfa 2b + ribavirin

INTERVENTIONS:
Drug: Celgosivir — 400mg qd + standard of care for 12 weeks
  Arms: 1
Drug: Celgosivir — 600mg qd + standard of care for 12 weeks
  Arms: 2
Drug: Peginterferon alfa 2b + ribavirin — Standard of care for 12 weeks
  Arms: 3

SUMMARY:
The objective of this study is to undertake an initial evaluation of the safety, tolerability, antiviral effect, and pharmacokinetics of celgosivir in combination with peginterferon alfa-2b and ribavirin in patients with chronic HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age, inclusive
* primary diagnosis of chronic HCV infection, genotype 1
* Interferon-based treatment-naïve
* Body Mass Index of 18 to 30, inclusive

Exclusion Criteria:

* patients previously treated with Interferon-based therapy
* patients with diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Safety analysis | 12 weeks
HCV viral load | 12 weeks
Pharmacokinetics of celgosivir/castanospermine | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jim Pankovich, Study Director — BioWest Therapeutics Inc
Locations (3):
- Canada (3):
  - Liver and Intestinal Research Centre, Vancouver, British Columbia
  - Cantest, Vancouver, British Columbia
  - Biovail Contract Research, Toronto, Ontario